CLINICAL TRIAL: NCT04011800
Title: Catheter Ablation vs. Antiarrhythmic Drugs and Risk Factor Modification. PRAGUE-25 Randomized Study
Brief Title: PRAGUE-25 Trial. Catheter Ablation vs. AADs and Risk Factor Modification.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: General Teaching Hospital, Prague (Other); Brno University Hospital (Other); Hospital Podlesi (Other); Regional Hospital Liberec (Other)
Responsible Party: Principal Investigator, Pavel Osmancik, head of the department of cardiac arrhythmias, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRAGUE-25
Record Dates: First submitted 2019-06-28; First posted 2019-07-09 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; risk factor modification
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: Patient will be randomized into catheter ablation (CA) arm or AADs and risk factor modification (RFM) arm
Masking Description: prospective, randomized, open - label, non-inferiority study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catheter ablation (Active Comparator): Patients will undergo catheter ablation of atrial fibrillation.
  Interventions: Procedure: Catheter ablation
- Risk factor modification (Experimental): Patiemt will undergo risk factor intervention and antiarrhythmic drugs
  Interventions: Combination Product: Risk Factor Modification

INTERVENTIONS:
Procedure: Catheter ablation — Pulmonary vein isolation, or additional left or right-sided atrial lesions.
  Arms: Catheter ablation
Combination Product: Risk Factor Modification — dietary restriction, physical exercise, reduced alcohol intake with antiarrhythmic drugs
  Arms: Risk factor modification

SUMMARY:
Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia with a prevalence of 2% in general population. Incidence and prevalence of AF has been slightly increasing due to increasing age, improved ability to treat cardiac diseases, and higher incidence of obesity and other risk factors associated with AF. AF is associated with higher morbidity and mortality mainly caused by heart failure and stroke. Catheter ablation (with pulmonary vein isolation as a cornerstone) presents the most effective treatment method of AF. Recent observational studies have shown that intensive risk factor and lifestyle modifications, such as weight loss, reduced alcohol intake, and increased physical activity, are also associated with improved rhythm outocome. Head-to-head comparison of this very different methods has not been done yet. The aim of the project is to compare the effect of catheter ablation with lifestyle modification (risk factor modification) in a prospective, randomized, multicenter study on the maintenance of sinus rhythm (monitored using implantable ECG reveal), and on the progression of the fibrosis of the left ventricle.

DETAILED DESCRIPTION:
GOALS OF THE PROJECT The aim of our study is to compare the effect of the invasive strategy (catheter ablation) of atrial fibrillation with non-invasive strategy (non-amiodarone antiarrhythmic drugs with risk factor modification) in a prospective, multicenter, randomized, non-inferiority study. The main hypothesis is that strict risk factor modification (weight loss, physical exercise improvement, and alcohol reduction) with AADs in patients with AF will be associated with similar rhythm outcomes as catheter ablation. Beside the AF-recurrence as the primary endpoint, the secondary endpoints will be the AF burden (assessed using repeated Holter recordings), change in cardiorespiratory exercise (assessed using cardiopulmonary exercise test), MRI endpoints (diffuse myocardial fibrosis, epicardial adipose tissue), QoL (assessed using specific questionaiires), and metabolic endpoints (lipids, pro-inflammatory cytokines),

JUSTIFICATION OF THE PROJECT The main reason for the project is the large and ever-increasing number of AF patients, especially in light of the significant incidence of obesity in AF patients. Keeping in mind the high number of AF patients (≈ 2% of the population), its increasing incidence and prevalence, even if CAs were associated with a 100% success rate, it would be impossible to treat all AF patients using CA. A significant portion of patients with AF are obese. For instance, the median BMI was 29.2 in the EAST-AFNET Trial and 30 in the CABANA Trial. Furthermore, and this is the second reason for the project, a significant portion of AF patients are afraid of invasive procedures and would prefer a noninvasive approach if the efficacy of this approach is known. The third reason is to compare the effect of these two different methods on the structural and metabolic abnormalities associated with AF and obesity

METHODS The study is planned as prospective, multicenter, randomized, non-inferiority trial comparing two different approaches in the treatment of AF. Symptomatic AF patients indicated for rhythm control strategy (i.e. restoriation and maintenance of SR) will be enrolled and randomized to catheter ablation or risk factor modification.

Study population - inclusion criteria (all of three have to be met for enrollment) (i) symptomatic AF (paroxysmal, persistent, or long-standing persistent), and (ii) BMI ≥ 30, and (iii) signed informed content

Study population - exclusion criteria:

* permanent AF
* severe valve disease (significant aortic stenosis, mitral regurgitation ≥ 3)
* left ventricular ejection fraction < 40%
* severe pulmonary hypertension (PAP > 40 mm Hg)
* history of tachycardia-induced cardiomyopathy
* planned revascularization
* pregnancy
* left atrial size ≥ 60 mm
* BMI less than 30, or BMI ≥ 40
* indication for surgical treatment of obesity
* age ≥ 75 let
* a significant physical limitation that could affect physical activity (musculoskeletal disorders, COPD)
* life expectancy less than 2 years Patients with significant structural heart disease (left ventricular dysfunction, significant valve disease, moderate or severe pulmonary hypertension, significant left atrial dilation) will be excluded. Also, patients who could not actively participate (musculoskeletal disorders, heart failure, patients older than 75 years) in regular physical activity will be excluded. Diabetes will be an exclusion criterion because of significant interference associated with antidiabetic medication relative to some of the endpoints.

BASELINE DIAGNOSTIC EXAMINATION After informed content is given, all patients will undergo baseline anthropometric measurements and baseline examinations. It will include (1) baseline evaluation of physical fitness - functional diagnostic, (2) echocardiography, (3) quality of life analysis, (4) blood biochemistry and cytokine analysis, and (5) a baseline one-week ECG Holter recording, (6) cardiac MRI. All these examinations will be done within four weeks after randomization.

Functional diagnostic (anthropometric measurement and cardiopulmonary exercise test) After enrollment, standard anthropometric measurements will be gathered, i.e., height, weight, percentage of body fat, and waist-to-hip ratio measurements. Functional diagnostics will be performed in all patients. Based on the results of functional diagnostics, an individualized and optimized physical training program will be prepared in patients randomized to the RFM arm.

An initial maximum symptom limited cardiopulmonary exercise test (CEPT) will be carried out within one month of enrollment.

Cardiac magnetic resonance (CMR) CMR will be done using 1.5 Tesla scanners located at each of the three participating centers. Before CMR evaluation, the ventricular rate will be optimized with a target ventricular rate < 100/min.

RANDOMIZATION Patients will be randomized to the catheter ablation group (CA) or risk factor modification group plus AADs (RFM) in a 1:1 ratio; randomization will be done using randomization software that will account for age, initial BMI, and AF type, with the goal of having comparable groups relative to those characteristics. The randomization process will be done outside all participating centers.

TREEATMENTS A. Catheter ablation (CA) arm CA will be done within two months of randomization. In patients with paroxysmal AF, a PVI will be performed. In patients with non-paroxysmal AF forms, additional lesion sets, except for a PVI, will be allowed according to the practice of each participating center. The CA will be done using a 3D mapping system, intracardiac echocardiography, contact-force sensing ablation catheters, and ablation index to achieve the maximum available safety and to allow for the delivery of maximally effective ablation lesions. During the study course, several centers have started to prefer pulsed-field ablation. Per amendment, pentaspline pulsed-field ablation catheter with corresponding pulsed-field energy generator can be used for catheter abaltion. Similarly as with radiofrequency ablation, the goal will be to effectivelly isolate pulmonary vein. Based on the discretion of the operator, additional lesions could be done.

The first three months following catheter ablation will be considered as a "blanking period," i.e., AF reoccurrences won´t be assessed as an endpoint. If AF reoccurs during this period, treatment using AADs or cardioversion will be allowed. Three months after ablation, AADs will be discontinued.

B. Risk factor modification and antiarrhythmic drugs arm (RFM arm)

The aim will be (1) a 10% weight loss over 6-12 months,(2) an increase in physical fitness, and (3) a reduction in alcohol consumption. Nutritional intervention: the initial patient consultations with nutritional specialists will be done during the first month after enrollment. A low-calorie, high protein, and low glycemic index dietary menu will be suggested and optimized by a nutritional specialist for each patient. Patients will have regular consultations with dietary specialists at least once a month during in-person visits in the early follow-up or by phone visits later during the follow-up; however, non-planned dietary consultations will be available every working day by calling a dietary specialist or using mobile application. Moreover, patients will be encouraged to record the calory intake in the OBEFIS application (either on the web www.obefis.cz, or using the mobile application) on a daily basis, and the recordings will be discussed during the visits with dietary specialists.

All patients will have an initial consultation with a physiotherapist (after the CPET) to set the type and intensity of the physical intervention. The recommended physical intervention will consist of three types of activities: (1) regular gym-based training (in small groups or individual training with trainer),(2i) individual aerobic training (fast walking or similar aerobic activity), and (3) home-based training: 20 min physical exercise sets. The type and ratio of the aforementioned physical exercises will be changed over the study period. In the first three months, there will be more emphasis on regular gym-based training under surveillance. The goal will be to teach patients how to properly perform all the exercises as well as assisting patients in getting used to regular exercise. At the end of the third month, the majority of patients should be accustomed to regular physical activity; the ratio of types of physical activities will be changed to a greater emphasis on individual physical activity. However, based on the patient´s experiences with physical activity in the past, and their options regarding participation in the organized training, activities will be individualized, and some patients may start the physical activity program individually without previous participation in group-based or surveillance-based training.

The intensity and frequency will be set individually based on initial CPET. The ESC guidelines for obese individuals recommend that a minimum of 150 min/week of moderate-intensity endurance exercise training should be combined with three weekly sessions of resistance exercise with the heart rate during the activity being 55-74% of the maximum HR (31). As such, the physical intervention will be based on regular (mainly moderate, ~ 55-74% of the maximum HR) intensity aerobic exercise that will be gradually increased from 60 min/week up to 200 min/week (in some individuals up to 300 min/week), and then continued until the end of the study. Patients will be taught how to use their optimal heart rate for aerobic exercise; for moderate-intensity training, the heart rate during the activity should be 55-74% of the max. HR. They will also be warned about exceeding their maximum possible heart rate (i.e., not exceeding 85% of the maximum heart rate). Since it is known that the adherence of patients to regular activity is affected by activity monitoring, all patients will have an opportunity to be monitored during each exercise using remote heart rate monitoring (fitness bands) and the OBEFIS smartphone application. It also allows monitoring of the heart rate during activity and an online discussion with therapists during the follow-up period.

For patients in the RFM arm, contrary to patients in the CA arm, non-amiodarone AADs will be allowed during the whole study period. The reoccurrence as AF/AT as an endpoint will be considered starting at the 6-month visit, including a 7-day Holter, which is scheduled to be done at the 6-month visit.

In both arms, in case of a reoccurrence of symptomatic AF or atrial tachycardia (AT), re-do ablations, cardioversion, or AADs treatment during the follow-up period will be allowed in accordance with the current guidelines and practices of participating centers. However, because the indication for the aforementioned procedures or AAD initiation will be a reoccurrence of AF or AT, it will be assessed as the primary endpoint (i.e., AF reoccurrence).

OUTPATIENT FOLLOW-UP The follow-up protocol and ECG monitoring will be similar for both arms. Starting on the day of the catheter ablation (D0 in the ablation arm), or at the start of the metabolic activity (D0 in the RFM arm, approx. 3-4 weeks after randomization), follow-up visits will be scheduled at 3, 6, 9, and 12 months during the first year, and then every six months. At the 3-month follow-up visit, patients in AF (from both groups) will undergo electrical cardioversion.

A routine 12-lead ECG will be recorded at each follow-up visit, along with a physical examination of the patient and a medical history update. Long-term ECG recording will be done using a 7-day Holter recording at baseline, and then at the 6, 9, and 12 months visits during the first year, and then every six months in the second and third years. Baseline 7-day ECG Holter recordings will be done in all patients after enrollment and within the first three weeks for patients on antiarrhythmics before study entry; this will serve as background for comparisons of AF burden.

The first three months in the CA arm and the first six months in the RFM arm will serve the blanking period. Starting at 3M (CA) or 6 M control (RFM) control, any reoccurrence of AF/AT will be considered an endpoint.

At the 12-month follow-up visit, echocardiography, MRI examination, anthropometric measurements, and CPET will be done. Blood will be drawn for cytokine analysis, and patients will also be asked to complete follow-up QoL questionnaires.

ENDPOINT MONITORING The AF reoccurrence will be detected either using planned 7-day Holter recordings (at the 6, 9, and 12 m visits), during all planned outpatient visits using a standard 12-lead ECG, and any time during the follow-up at an emergency non-planned visit also using a standard 12-lead ECG (starting at the three-month visit in the CA arm and the six-month visit in the RFM arm). The occurrence of AF > 30 sec during planned 7-day Holter recordings, either planned or emergency, a non-planned visit will be assessed as a primary endpoint. Importantly, during all outpatient in-person visits, AF reoccurrence has to be documented using an ECG (i.e., a patient´s description of "palpitations" without ECG evidence will not be assessed as AF reoccurrence).

STUDY OUTCOMES

Primary endpoints:

1) AF reoccurrence (any AF or atrial tachycardia lasting more than 30 sec) SECONDARY OUTCOMES

1. AF burden: calculated using all Holter recordings as a percentage of time spent in AF or AT
2. AF reoccurrence and AF burden at the 12-month visit
3. Hospitalization for AF reoccurrence and/or emergency room visit due to AF
4. A composite of stroke, cardiovascular death, or hospitalization for heart failure
5. Changes in QoL questionnaires between baseline and 12 months
6. Change in cardiorespiratory fitness as assessed using CPET between baseline and 12 months (ml/kg/min)
7. Metabolic endpoint: changes in weight, fasting glucose, lipid levels, glycated hemoglobin, and cytokines associated with inflammation and atrial function (interleukin-6, natriuretic peptides)
8. Imaging endpoints: change in the amoubnt of EAT and % in ventricular fibrosis between baseline and the 12-month examination (MRI), and a change in left atrial parameters (echocardiography)

Power calculation and statistical analysis The expected efficacy of the Catheter ablation In a meta-analysis of RCT comparing CA with AADs, the single procedure success rate of CA OFF AADs was 57% (96%CI 50-64%) In the CABANA trial, AF freedom was present in 63.6% of the ablation patients by 12 months. The expected one-year AF freedom in the CA arm is ≈ 60%.

The expected efficacy of AADs and RFM In a meta-analysis of 24 randomized control trials comparing AADs with placebo, the overall success rate of AADs, defined as the disappearance of arrhythmia during follow-up, was present in 52% (95%CI 47%-57%) of patients on AADs. The highest efficacy was achieved using amiodarone (58%), followed by flecainide and propafenone (48%). In the CABANA trial, by 12 months, the one-year AF freedom on AADs was present in 47.1% of patients. Finally, in the recently published STOP-AF trial, one-year AF freedom (assessed using repeated 24-Hour Holter recordings) was present in 45.0% (95%CI 34.6-54.7) of patients, but only 2% were on amiodarone, and the rest were on flecainide, sotalol and propafenone. Therefore, a one-year AF freedom of 45% could be expected for non-amiodarone AADs. In the LEGACY study, the achieved AF freedom significantly depended on weight loss. Relative to weight loss, patients were categorized as >10%, 3%-9%, and < 3% weight loss. During follow-up, 45.5% patients in the >10%, 22.2% in the 3-9%, and 13.4% in the < 3% group remained AF-free without AADs or ablation. In the ARREST AF, at the final follow-up (mean duration 41 months), 32.9% of patients in the RFM arm vs. 9.7% controls remained AF-free after a single CA procedure. No study has compared the additive effect of weight loss on top of AADs; however, an additional effect of 20% could be expected in these patients. Therefore, we expected a ≈ 65% one-year AF freedom in the noninvasive treated patients.

According to the aforementioned data, we expect one-year AF freedom in 65% of patients in the RFM arm and 60% in the CA arm. The primary analysis will be done using the intention-to-treat principle; however, based on the non-inferiority nature of the study, a per-protocol analysis will be done. The sample size calculation assumed: 80% power, 5% one-sided alpha, a non-inferiority margin of 12% (or 1.65, if expressed as an odds ratio). Using this assumption, 202 patients (101 in each arm) will need to be enrolled to prove non-inferiority of the noninvasive arm relative to the invasive arm. With an expected drop-out rate of 5%, therefore, 212 patients will be enrolled.

Study organization, randomization process and data management

The institution responsible for the organization and implementation of the study is the 3rd Faculty of Medicine, Charles University in Prague, Czech Republic. Data obtained during each patient visit will be collected using a safe electronic CRF form. A tailor-made website was developed for the study. Each participating medical center will have access to a dedicated part of the website. The database and randomization software has been prepared by an outside party (i.e., the Institute of Biostatistics and Analyses, Masaryk University, Brno, Czech Republic), and no investigator will have access to the database or the randomization software.

Safety and endpoint monitoring The local investigator at each site will continuously review safety data during the trial. A Data Safety Monitoring Board (DSMB) will be constituted before the commencement of the trial. Reporting of adverse events will be reported to the DSMB immediately by the principal investigator. Serious adverse events (SAE) will be defined as life-threatening events or events resulting in death or hospitalization. All SAEs linked with the study will be reported to the DSMB, to the FNKV Ethics Committee (a multicenter ethics committee, EC), and to the local ECs within 24 hours of study staff becoming aware of the event. Clinical endpoints will be analyzed by a dedicated clinical endpoint committee. The recording and analyses of all Holter recordings in all participating centers will be done centrally using an MDT (medical data transfer) company.

DISCUSSION In the last five years, lifestyle modification with risk factor management has been shown to be a very promising treatment modality for AF. AF is the most common sustained cardiac arrhythmia, with an estimated worldwide prevalence of about 33.5 million people. According to recent epidemiological studies, its prevalence may triple by 2050 Even if catheter ablations were associated with a 100% success rate, it would be impossible to treat the current or projected numbers using catheter ablations. Furthermore, a substantial number of patients would prefer a non-invasive treatment if both strategies were comparable. So while risk factor modification studies may seem to offer a panacea, those studies suffer from significant limitations and possible biases. For example, the most important and most extensive studies were both non-randomized, and all patients had either a history of catheter ablation (ARREST-AF) or were without a history of catheter ablation, but catheter ablation was allowed without limitations, based on the judgment of the attending physician during the follow-up period (LEGACY). A randomized study that directly compares catheter ablation with a modern noninvasive strategy has yet to be done. If the effect of both strategies were comparable, the noninvasive strategy could be offered to patients with a preference for a noninvasive treatment. Only a randomized study can really answer the question of how effective lifestyle modification is supported by safe non-amiodarone AADs compared to a modern invasive strategy. Additionally, a randomized study has the potential to show the additional effect of both strategies (effect on CMR measures or pro-inflammatory cytokines concentrations) and to determine which patients would most likely benefit from a non-invasive treatment, thus increasing the number of successfully treated AF patients, without the use of invasive methods.

ELIGIBILITY:
Inclusion Criteria (all three must be met):

* symptomatic atrial fibrillation
* BMI ≥ 30, and
* signed informed content

Exclusion Criteria:

* permanent AF
* severe valve disease (significant aortic stenosis, mitral regurgitation ≥ 3)
* left ventricular ejection fraction < 40%
* severe pulmonary hypertension (PAP > 40 mm Hg)
* history of tachycardia-induced cardiomyopathy
* manifest coronary artery disease
* pregnancy
* left atrial size ≥ 60 mm
* indication for surgical treatment of obesity
* BMI ≥ 40
* diabetes mellitus on insulintreatment
* age ≥ 75 let
* a significant physical limitation that could affect physical activity (musculoskeletal disorders, COPD)
* life expectancy less than 2 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Freeedom from atrial fibrillation and/or atrial tachycardia | 6 months after the procedure at least, and later during the follow-up
  An absence of any paroxysm of atrial fibrillaton or atrial tachycardia lasting then 30 second, as assessed using repeated 7-day Holter recordings

SECONDARY OUTCOMES:
AF burden | baseline, than 6,9,12m and every 6 months
  The percent of time spending in atrial fibrillation or atrial arrhythmia, as assessed using repeated 7-day Holter recordings
Hospitalization for AF | 12 months
  The number of hospitalizations or emergency visits due AF
A composite of stroke, cardiovascular death, or hospitalization for heart failure | 12 months
  Clinical endpoint, composite number of events associated with AF
MRI endpoint | baselien and 12months
  Change in the amount of epicardial adipose tissue(ml) and in the ventricular myocardial fibrosis (%)
Change in cardiorespiratory fitnes | baseline and at 12 months
  Change in cardiorespiratory fitnes assessed using exercise test (ml/kg/min)
Changes in QoL questionnaires between baseline and 1 year | 12 months
  Change in quality of life, assessed by specific questionnaire in one year
Weight | 12 months
  Change in weight between between baseline and 12 month level
Fasting glucose | 12 months
  Change in fasting glucose between baseline and 12 month level
Triglycerides | 12 months
  Change in trigylcerides between baseline and 12 month level
Interleukin-6 | 12 months
  Change in interleukin-6 concentration between baseline and 12 month level

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiocenter, 3rd Medical School, Charles University and University Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
The primary analysis is planned after 6 monts of follow-up of the last enrolled patients. After that, an extension of follow-up for three additional years is planned according to the protocol. Study data will be shared when the follow-up extension is finished and analyzed. Data will be available upon reasonable request. Deidentified patient data will be stored at the Institute of Biostatistics and Analyses, Masaryk University, Brno, Czech Republic, and will be available after request to principal investigator for further analyses and meta-analyses.
Supporting Information: CSR, Analytic Code
Time Frame: Three years after the end of follow-up, data will be available
Access Criteria: upon a request to the principal investigator. Only for the purpose of additional analyses - subanalysis or meta-analysis with similar trials.

REFERENCES:
- [Derived] Osmancik P, Havranek S, Bulkova V, Chovancik J, Roubicek T, Herman D, Carna Z, Tuka V, Matoulek M, Fiala M, Jiravsky O, Stregl-Hruskova S, Latinak A, Kotryova J, Jarkovsky J. Catheter ablation versus antiarrhythmic drugs with risk factor modification for treatment of atrial fibrillation: a protocol of a randomised controlled trial (PRAGUE-25 trial). BMJ Open. 2022 Jun 15;12(6):e056522. doi: 10.1136/bmjopen-2021-056522. PMID 35705334